CLINICAL TRIAL: NCT05961878
Title: Efficacy of Diet in Elderly With Type 2 Diabetes
Brief Title: Diet in Elderly With Type 2 Diabetes
Acronym: SARC-OLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Emanuela Orsi, medical doctor, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sarcopenia-diabetes
Record Dates: First submitted 2023-07-06; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Sarcopenia; Sarcopenic Obesity; Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Complications
MeSH Terms: conditions — Sarcopenia; Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Complications | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sarcopenic (Experimental): subjects with sarcopenia diagnosis
  Interventions: Dietary Supplement: mediterranean diet with adequate protein intake
- Non sarcopenic (Placebo Comparator): subjects without sarcopenia diagnosis
  Interventions: Dietary Supplement: mediterranean diet with adequate protein intake

INTERVENTIONS:
Dietary Supplement: mediterranean diet with adequate protein intake — balanced mediterranean diet with 1.1 g/kg die protein intake

SUMMARY:
Sarcopenia is characterized by progressive and generalized loss of skeletal muscle mass which may affect performance. Diabetes can affect muscle cell function, making sarcopenia worse.

This is a prospective and interventional study on a elderly population affected by type 2 diabetes mellitus. All subjects, recruited will undergo tests for the diagnosis of sarcopenia according to the EWGSOP2 criteria. All subjects, both sarcopenic and non-sarcopenic, will be introduced to a targeted nutritional program aimed at improving the composition of the diet, in terms of both micro- and macro-nutrients.

DETAILED DESCRIPTION:
The sample will consist of about 100 subjects (50 sarcopenic and 50 non-sarcopenic) who receive the nutritional program. Particular attention will be paid to the intake of an adequate protein intake for the elderly subject (1.1 g/kg/day). A food diary will be required to assess daily protein-calorie intake and questionnaires to assess daily physical activity and quality of life.

The primary objective is to assess the efficacy of nutritional intervention in elderly affected by type 2 diabetes mellitus and sarcopenia. The secondary objective is to identify the prevalence of sarcopenia in patients with type 2 diabetes mellitus compared to non-diabetic subjects and to verify the relationship between pharmacological therapy and the presence of sarcopenia as well as evaluate any changes in style and quality of life and of glycometabolic compensation.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* BMI >20 kg/m2
* HbA1c ≥6.5% (48 mmol/mol) e ≤10% (86 mmol/mol)

Exclusion Criteria:

* T1DM or LADA
* Patients with serious primary diseases of heart, brain, liver, kidney and hematopoietic system

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-31 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Handgrip test | 1 years
  Increase of hand grip strength (units: kg)

SECONDARY OUTCOMES:
Glycemic control | 1 year
  HbA1c (units: mmol/mol)
Anthropometric parameters: BIOIMPEDENTIOMETRIC PARAMETERS | 1 year
  fat mass and free fat mass (units: % of total mass)
Dietary lifestyle | 1 year
  variations in intake of simple sugars, animal protein rich foods, saturated fats and cholesterol, UDM: grams/die. All the informations will be collected using 5days food diaries, completed by the patients

OTHER OUTCOMES:
health-related quality of life | 1 year
  assesed Sacopenia Quality of life (SarQoL)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy